CLINICAL TRIAL: NCT03626389
Title: Clinical Course and Prognostic Factors of Patients Receiving Physiotherapy Services in Primary Health Care in Norway (FYSIOPRIM)
Brief Title: Clinical Course of Patients Receiving Physiotherapy Services in Primary Health Care
Acronym: FYSIOPRIM
Status: Completed | Type: Observational
Sponsor: University of Oslo (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other); Norwegian University of Science and Technology (Other); Trondheim Kommune (Other)
Responsible Party: Principal Investigator, Nina K. Vollestad, Professor, University of Oslo
Other Study IDs: FYSIOPRIM
Record Dates: First submitted 2018-06-18; First posted 2018-08-13 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Musculoskeletal Diseases or Conditions; Neurologic Disorder; Widespread Chronic Pain; Psychosomatic Disorder; Arthritis; Injuries
Keywords: physiotherapy; primary health care setting
MeSH Terms: conditions — Musculoskeletal Diseases; Nervous System Diseases; Chronic Pain; Psychophysiologic Disorders; Arthritis; Wounds and Injuries | interventions — Physical Therapy Modalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving physiotherapy in primary care: Physiotherapy, without predetermined selection of specific modalities
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Physiotherapy

SUMMARY:
Background: Physiotherapists (PTs) in primary health care manage patients with a large variation in medical diagnosis, age, functional status, disability and prognosis. Lack of knowledge and systematically collected data about patients treated by PTs in primary health care has prompted this longitudinal observational physiotherapy project in Norway. This paper aims to describe a method for developing a database of patients managed by PTs in primary health care to study patients' characteristics, treatment courses and prognostic factors.

The study is a longitudinal observational project, following patients through physiotherapy treatment periods in primary health care in Norway and until one year after inclusion. The project involves both private practice and municipally employed PTs working in primary health care in eight municipalities in Norway. The participants are recruited to three different parts of the project depending on age and whether they are referred to a private practice or a municipally employed PT. All data are recorded electronically, transferred and stored securely. All patients complete extensive questionnaires providing information about demographics, disability and function, pain related variables, treatment and evaluation of treatment as well as clinical tests. The PTs have access to their own patients' data. The investigators have also prepared for linkage to national patient registers and population-based studies to be able to gather further important data.

This project will have important implications for physiotherapy services in primary health care. The database already contains almost 3000 patients, and data collection is ongoing. Preliminary analyses suggest that the patients included so far are representative of the larger population of patients treated by private practice or municipally employed PTs in Norway. This large scale prospective physiotherapy project will provide knowledge about the patient groups treated, treatment given as well as short and long term outcome of the patients.

DETAILED DESCRIPTION:
The primary aim of the FYSIOPRIM project is to build a database by systematically collecting data from baseline throughout the intervention period and beyond, including both patient-reported outcome measures, the patients' and PTs' goals and plans for intervention, and their evaluation thereof. This will enable description of patients receiving physiotherapy services, of goal-setting and type of interventions and how general health, physical function and relevant clinical factors change throughout and after a treatment period. Secondly, the investigators want to study associations and interaction effects between and among clinical characteristics, interventions and change as well as perform health-economic evaluations. The investigators will also examine how physiotherapy practice is affected by using the system for systematic registration of clinical data and effects of such registration. Moreover, the investigators will be able to compare patients receiving physiotherapy services with information from national patient registries. In addition, elderly participants' physical fitness, balance and walking ability will be examined to study associations between these aspects of physical functioning and health-related quality of life, self-reported physical and psychological functioning as well as response to physical fitness tests. The investigators will compare data from this group of elderly with data from other patients with musculoskeletal complaints who receive physiotherapy treatment, and with similar data from large population-based studies in Norway. Finally, this project enables methodological studies to validate clinical tests and questionnaires.

Design and setting This is a longitudinal observational project following patients through physiotherapy treatment periods in primary health care in Norway and until one year after baseline. The project involves both private practice and municipally employed PTs working in primary health care in eight municipalities of Norway; Lørenskog, Ski, Nedre Eiker, Lillehammer, Stavanger, Bergen, Trondheim and Alta. All five health regions of Norway are represented. The Norwegian Health care system is publicly funded. PTs working as private practitioners have an agreement with the municipality. Hence, they are partly paid by the municipality (as a financial support for practice) and partly paid per visit by the Norwegian Health Economics Administration (HELFO) and the patient's charge (maximum around 200 Euro per patient per calendar year). Patients seeking physiotherapy services in private practice will normally meet at the PT's clinic.

Municipally employed PTs are on fixed salary. They work in an out-patient setting, and their patients receive physiotherapy services in their usual daily environment, i.e. for children at home, in kindergarten or in school, and for elderly patients often in their own home. There are no clear guidelines for which patients that should receive physiotherapy from a private practice or a municipally employed PT. The choice can be based on previous personal experiences with physiotherapy, the possibility to visit a clinic, evaluation of need and/or benefit of treating the patients in their own setting.

Characteristics of participants

The participants are recruited to three different parts of the project depending on age and whether they are referred to a private practice PT or to a municipally employed PT (in this project, these PTs are from Trondheim). The three parts of the project are:

1. Adults seeking physiotherapy services in private practice This part of the project started data collection in June 2015, and data collection is planned to continue through June 2020. From January 2016 through December 2017, data were collected from a total of 2754 patients above the age of 18 years seeking physiotherapy treatment from 111 PTs in eight municipalities in different parts of Norway, including 536 patients already in treatment. Among the 111 PTs, 78 (70.3%) are general PTs, 20 (18.0%) are manual therapists and13 (11.7%) are PTs with special education in psychomotor physiotherapy. Seventy-seven (69.4%) of the PTs are working in Trondheim.
2. Adults and elderly receiving physiotherapy services in Trondheim Municipality This part of the project collected data from the beginning of May 2016 to the end of May 2018. From January 2016 until the end of September 2017, data were collected from 684 adults and elderly patients receiving physiotherapy services from approximately 55 PTs working with adults and elderly in the municipality of Trondheim in Norway. Adults and elderly may be referred from general practitioners, occupational therapists, health professionals at health care centers, rehabilitation centers or hospitals, or by proxy. The physiotherapy services to adults and elderly include early intervention, activities of daily living (ADL) rehabilitation and ordinary physiotherapy, all of which are typically delivered in a home setting. Early intervention is a collaboration between health and welfare centers and units for physiotherapy and occupational services and is offered to patients in need of limited services who are referred to municipality health care services for the first time. ADL rehabilitation are offered to patients in risk of functional deterioration who are receiving home based services, while ordinary physiotherapy is offered to patients in need of more specific physiotherapy services.
3. Children receiving physiotherapy services in Trondheim Municipality This part of the project collected data from May 2016 through April 2017. During this period, data were collected from 165 children aged 0-18 years receiving physiotherapy services from approximately 25 PTs working with children in the municipality of Trondheim in Norway. For children, physiotherapy may be initiated on referral from parents, personnel at kindergarten or in school, general practitioners, occupational therapists, and health professionals at primary health care centers or hospitals. The children typically receive physiotherapy services at the primary health care centers, in their own home or in kindergarten or at school, depending on the child's usual primary location and condition.

Data collection Patients are asked to participate at their first time encounter with a physiotherapist in primary health care. Project information and consent forms are available in Norwegian and English. The investigators collect baseline data in two steps. First, the therapist and the participant together fill in information about the main problem, and jointly agree on goals for treatment and a treatment plan. The therapist also asks the participant for their own specific functional problem using the Patient-Specific Functional Scale (PSFS). The therapist provides information about the referral, diagnosis and whether any disease-specific questionnaires should be used for this participant. Secondly, the participant completes questionnaires themselves, either using an e-tablet or through a web-link sent by e-mail. A set of outcome data are common to all, and in addition disease-specific outcome measures are included for some common patient groups.

Approximately 1 month after baseline (for participants seeking PTs in private practice), or 2-3 months after baseline (for participants receiving physiotherapy from municipally employed PTs), the therapist and the participant together evaluate goal achievement and fulfilment of the treatment plan so far. They also adjust these when needed and the participant recompletes the PSFS. Three months (for private practice) or six months after baseline (for participants receiving physiotherapy from municipally employed PTs), the PT and the participant again evaluate goal achievement and fulfilments of the treatment plan. The participant then completes the same standardized questionnaires as at baseline. The same questionnaires are also completed 6 and 12 months after baseline by participants treated by PTs in private practice using a web-link sent by smartphone or e-mail. All participants treated by PTs in private practice receive reminders once a week, up to three times, by sms and e-mail if they have not answered the questionnaires.

All data are collected electronically using an application run on a tablet or through a web-link. The software is provided by Infopad AS (www.infopad.no). Immediately after the completion of the questionnaires all data are transferred to a backend secure server with in-memory encryption. The PTs have access to their own participants' data either through a web-site and/or by importing data into their electronic medical journal. The journal number of the participant is used as the study identifier to enable data flow between the electronic medical journal and the secure backend server. The data from all participants are copied to a secure server at the University of Oslo set up for research purposes (Services for Sensitive Data). Data management is done according to the quality assurance system of the University of Oslo. The investigators have prepared for linkage between data from FYSIOPRIM and data from national patient registers. This will be done by use of the participant's journal number to access their unique 11-digit Norwegian personal number.

All the data are collected electronically, thereby avoiding the possibility of mistakes when transferring data from paper forms to electronic data. Data management is performed using STATA 15 (Stata Corp., College Station, Texas, USA). The raw data are stored in a secure database where only researchers associated with the project have access. Before data can be used for analyses a range of automated procedures for data preparation and quality checking are performed using standardized, written scripts in STATA. Examples are to check, i) patterns of missing data, ii) values outside the possible range of a variable (e.g., age>120 years), iii) conflicting answers (e.g., pregnancy and male) and iv) unexpected frequency distributions for categorical variables. The investigators will explore each variable graphically using histograms and plots to evaluate the data distribution. Descriptive statistics will be used to describe the patient populations using parametric or non-parametric statistics according to the data distribution. Detailed descriptions of all the statistical analyses planned are beyond the length of this paper. Thus, specific analyses related to investigation of associations between variables, prognosis and clinical course will be described in future publications.

ELIGIBILITY:
Inclusion Criteria:

* any patient seeking or receiving physiotherapy services in primary health care

Exclusion Criteria:

* Not understanding Norwegian or English language

Ages: 0 Years to 125 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients are recruited through physiotherapists in primary health care.
Sampling Method: Non-Probability Sample
Enrollment: 4985 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Health-Related Quality of LIfe - assessed by EuroQual 5 Dimensions questionnaire (EQ-5D) | Baseline, 3, 6 and 12 months
  Utility measure of Health related quality of life. Range -0.59 (worst) to 1 (best)
Change in Patient-Specific Functional Scale (PSFS) | Baseline, 1, 3, 6 and 12 months
  Participants identify activities that are difficult to perform and scores them from 0 (cannot perform) to 10 (perform without problems)
General Perceived Effect | 3, 6 and 12 months
  A global assessment of change- 7 level scale. Score range 1 (very much better) to 5 (very much worse)
Change in Pain intensity | Baseline, 1, 3, 6 and 12 months
  Pain intensity assessed by a numeric rating scale. Range 0 (no pain) to 10 (worst imaginable)

SECONDARY OUTCOMES:
Change in Work participation | Baseline, 3, 6 and 12 months
  Sick leave (% of full time)
Change in work ability | Baseline, 3, 6 and 12 months
  One questeion. Range 0 (cannot work at all) -10 (can work at my very best)
Change in pain distribution | Baseline, 3, 6 and 12 months
  Participants marks pain distribution in a drawing- max no of sites:112
Change in use of analgesics containing paracetamol | Baseline, 3, 6 and 12 months
  Participants indicate if used last week and how often (less than daily, 1-4 per day, >5 per day)
Change in use of analgesics containing ibuprofen | Baseline, 3, 6 and 12 months
  Participants indicate if used last week and how often (less than daily, 1-4 per day, >5 per day)
Change in use of analgesics containing acetylsalicylacid | Baseline, 3, 6 and 12 months
  Participants indicate if used last week and how often (less than daily, 1-4 per day, >5 per day)
Change in emotional distress assessed by Hopkins Symptoms Check List (HSCL) | Baseline, 3, 6 and 12 months
  10 questions. Score range: 1 (best) to 4 (worst)
Change in Pain Self-efficacy | Baseline, 3, 6 and 12 months
  Pain Self-efficacy Questionnaire (2 items). Score range 0 worst) to12 (best)
Change in health related quality of life assessed by 15D | Baseline, 3, 6 and 12 months
  Utility merasure of Health related quality of life - range 0 (worst) to 1 (best)
Change in catastrophising thoughts assessed by Pain Catastrophizing Scale | Baseline, 3, 6 and 12 months
Change in Neck disability Index (NDI) | Baseline, 3, 6 and 12 months
  Questionnaire - Score range 0 (best) to 100 (worst)
Change in Oswestry Disability Index (ODI) | Baseline, 3, 6 and 12 months
  Questionnaire - Score range 0 (best) to 100 (worst)
Change in Shoulder Pain and Disability Index (SPADI) | Baseline, 3, 6 and 12 months
  Questionnaire for patients with shoulder pain - Range 0 (no disability) to 100 (completely disabled)
Change in Disability of the Arm, Shoulder and Hand score (Quick-DASH) | Baseline, 3, 6 and 12 months
  Questionnaire for patients with shoulder or arm pain - Range 0 (no disability) to 100 (completely disabled)
Change in temporal aspects of pain | Baseline, 3, 6 and 12 months
  Participants responds with yes/no to questions on continual pain and variability in pain intensity
Change in hip disability - assessed by the Hip Disability and Osteoarthritis Outcome Score (HOOS) | Baseline, 3, 6 and 12 months
  Hip disability questionnaire for patient with hip pain - 5 domains (pain, symptoms, ADL, sports/recreation, quality of life). Score range 0 (best) -100 (worst)
Change in pelvic girdle pain and disability assessed by the Pelvic Girdle Questionnaire | Baseline, 3, 6 and 12 months
  Quesionnaire questionnaire for patient with pelvic girdle pain - range 0 (no disability or pain) to 100 (high disability and pain)
Change in knee disability - assessed by the Knee Disability and Osteoarthritis Outcome Score (KOOS) | Baseline, 3, 6 and 12 months
  Knee disability questionnaire for patient with knee pain - 5 domains (pain, symptoms, ADL, sports/recreation, quality of life). Score range 0 (best) -100 (worst)
Change in physical functioning assessed by the Physcal function domain of Short Form 36 - (SF-36) | Baseline, 3, 6 and 12 months
  Sumscore with range 0 (worst) to 100 (best)
Change in insomnia problems assessed by the Insomnia Severity Index | Baseline, 3, 6 and 12 months
  Questionnaire - score range 0 (no insomnia problems) to 28 (severe insomnia problems)
Change in 6 min walk | Baseline, 3, 6 and 12 months
  6 min walk - timed measure (s)
Change in stair climb capacity | Baseline, 3, 6 and 12 months
  Stair climb 3 flights - up and down; timed measure (s)
Change in physical capacity assessed by 30 s sit to stand | Baseline, 3, 6 and 12 months
  Assessed as the number of times to complete a sit to stand and sit cycle witin 30 s
Short Physical Performance Battery | Baseline, 3, 6 and 12 months
  4 tests of Physical performance
Fulfilment of expectations | 3, 6 and 12 months
  One question
Benefit of treatment | 3, 6 and 12 months
  One question
Fulfillment of treatment goals | 3 months
  patients evaluate if the individually defined treatment goals are met, partially met or not met at all

CONTACTS AND LOCATIONS:
Overall Officials: Nina K Vøllestad, PhD, Principal Investigator — University of Oslo
Locations (2):
- Norway (2):
  - Approx 100 physiotherapists in Norway, Oslo
  - Physiotherapists in Trondheim, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
We plan to make the data available for other researchers. Anonymous data will be shared to all that asks and that provide a research plan approved by our steering committee. We will in principle be open for sharing all data, but we also need to verify that we comply with the approvals given. Deidentified data may be shared with other researchers given that they have secure storage and analytical platforms.
Time Frame: We plan to share data from 1 January 2019 and until our approval for use of data expires.
Access Criteria: Quality of proposal Scientific publication required as output to researchers Reports or white papers required as output to managers Financial support to carry out the project No conflict with ongoing research based on the data The use is in keeping with research ethical standards and regulations for use of personal data
URL: http://www.med.uio.no/helsam/english/research/groups/fysioprim/index.html

REFERENCES:
- [Derived] Handeland H, Evensen KAI, Robinson HS. Focus on physiotherapy and manual therapy for infants in Norway, a cross-sectional study on referral practice, and planned interventions. BMC Pediatr. 2025 Apr 9;25(1):282. doi: 10.1186/s12887-025-05627-3. PMID 40205420
- [Derived] Unsgaard-Tondel M, Vasseljen O, Nilsen TIL, Myhre G, Robinson HS, Meisingset I. Prognostic ability of STarT Back Screening Tool combined with work-related factors in patients with low back pain in primary care: a prospective study. BMJ Open. 2021 Jun 3;11(6):e046446. doi: 10.1136/bmjopen-2020-046446. PMID 34083340
- [Derived] Amundsen O, Vollestad NK, Meisingset I, Robinson HS. Associations between treatment goals, patient characteristics, and outcome measures for patients with musculoskeletal disorders in physiotherapy practice. BMC Musculoskelet Disord. 2021 Feb 13;22(1):182. doi: 10.1186/s12891-021-04048-4. PMID 33583404
- [Derived] Evensen KAI, Sellaeg S, Straete AC, Hansen AE, Meisingset I. Profile of children referred to primary health care physiotherapy: a longitudinal observational study in Norway. BMC Health Serv Res. 2021 Jan 6;21(1):16. doi: 10.1186/s12913-020-05988-8. PMID 33407440
- [Derived] Evensen KAI, Robinson HS, Meisingset I, Woodhouse A, Thielemann M, Bjorbaekmo WS, Myhre G, Hansen AE, Vasseljen O, Vollestad NK. Characteristics, course and outcome of patients receiving physiotherapy in primary health care in Norway: design of a longitudinal observational project. BMC Health Serv Res. 2018 Dec 4;18(1):936. doi: 10.1186/s12913-018-3729-y. PMID 30514287